CLINICAL TRIAL: NCT05716880
Title: FORMA - a Multicenter Randomized-controlled Trial to Evaluate the Efficacy and Safety of Ketoanalogues of Essential Amino Acids in Prophylaxis of Protein-energy Wasting in Nephrotic Syndrome
Brief Title: Ketoanalogues for Muscle Mass Loss in Nephrotic Syndrome
Acronym: FORMA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Collaborators: Medical University of Lodz (Other); Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ABM/FORMA/2021; 2022-000529-26 (EudraCT Number); 2021/ABM/01/00036-00 (Other Grant/Funding Number: Medical Research Agency, Poland)
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Nephrotic Syndrome
Keywords: nephrotic syndrome; protein-energy wasting; neph-PEW; lean tissue mass; Ketosteril; ketoanalogues
MeSH Terms: conditions — Nephrotic Syndrome | interventions — ketosteril

STUDY DESIGN:
Intervention Model Description: Randomization in 1:1 ratio with stratification by the type of glomerular disease (podocytopathy versus other type) and investigational site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KA+MPD (Experimental): Ketosteril + Medium Protein Diet (MPD) for 12 months
  Interventions: Drug: Ketosteril; Other: Medium Protein Diet (MPD)
- MPD (Active Comparator): Medium Protein Diet (MPD) for 12 months
  Interventions: Other: Medium Protein Diet (MPD)

INTERVENTIONS:
Drug: Ketosteril — Daily dose = 1 tabl / 5 kg of ideal body weight
  Arms: KA+MPD
Other: Medium Protein Diet (MPD) — MPD: daily protein intake of 0.8-1.0 g/kg of ideal body weight + up to 5 g based on daily proteinuria

SUMMARY:
The goal of this non-commercial clinical trial is to assess efficacy and safety of ketoanalogues of essential amino acids in the prevention of protein-energy wasting in nephrotic syndrome.

DETAILED DESCRIPTION:
Adult patients with new diagnosis or relapse of nephrotic syndrome and glomerular filtration rate of ≥ 30 mL/min/1.73m2 will be included in the study. Exclusion criteria will be a secondary cause of nephrotic syndrome, morbid obesity and severe diseases affecting nutritional status.

Participants will be randomly assigned to the intervention group (KA+MPD) or control group (MPD); randomization will be stratified by type of glomerular disease (podocytopathy or other type) and investigational site. The control group will follow the diet recommended in nephrotic syndrome - a medium protein diet (MPD) - under the care of a dietitian. Intervention group will receive Ketosteril (1 tablet for every 5 kg of ideal body weight) as an addition to the diet. All patients will also receive treatment for underlying glomerular disease in accordance with current guidelines and local practice.

The main objective is to assess the efficacy of Ketosteril as an add-on therapy in preventing the loss of lean tissue mass (LTM) over 6 months compared to a standard diet.

The additional aims include the assessment of muscle function parameters, nephrotic syndrome severity and laboratory indicators of catabolism.

ELIGIBILITY:
Inclusion Criteria:

* Nephrotic syndrome with serum albumin < 3.0 g/dL and daily proteinuria of > 3.5 g/day or > 50 mg/kg;
* New diagnosis or relapse of nephrotic syndrome (defined as: proteinuria of < 2.0 g/day or uPCR < 2000 mg/g in the last 6 months prior to relapse and prednison dose equal to or less than 10 mg/day in the last 3 months prior relapse);
* Glomerular filtration rate qual to or higher than 30 mL/min/1.73m2 based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

Exclusion Criteria:

* Diabetic kidney disease;
* Small vessels vasculitis;
* Systemic lupus erythematosus;
* Positive antinuclear antibodies, anti-dsDNA or antineutrophil cytoplasmic antibodies (ANCA);
* Positive anti-HIV or anti-hepatitis C antibodies, HBsAg;
* HbA1c >7%;
* Monoclonal gammopathy;
* Pregnancy;
* Body mass index >= 40 kg/m2;
* Severe acute or chronic disease affecting nutritional status;
* Neoplasm;
* Contraindication to Ketosteril;
* Alcohol or drug abuse;
* Mental disorders;
* Failure to comply with medical recommendations, lack of cooperation;
* Participation in other clinical trial or the use of Ketosteril in the last 1 year prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximum loss of lean tissue mass | 6 months
  The difference between the initial lean tissue mass (LTM) and the lowest LTM measured within 6 months, expressed in percentage. The non-inferiority hypothesis of Ketosteril use will be tested as the primary endpoint.
  LTM will be measured with bioimpedance spectroscopy.

SECONDARY OUTCOMES:
Maximum loss of lean tissue mass | 6 months
  The difference between the initial lean tissue mass (LTM) and the lowest LTM measured within 6 months, expressed in percentage. The superiority hypothesis of Ketosteril use will be tested as the secondary endpoint.
Neph-PEW diagnosis | 6 months
  The percentage of patients meeting criteria of nephrotic syndrome-associated protein-energy wasting (neph-PEW): reduction of LTM by 3% within 3 months or by 5% within 6 months.
6-minute walk test distance | 6 months
  Change in distance walked in the 6-minute walk test from baseline value; expressed in meters.
Handgrip strength (HGS) | 6 months
  Change in HGS value from baseline; expressed in kg.
Serum albumin | 6 months
  Change in serum albumin level from baseline value; expressed in g/dL.
Urinary protein/creatinine ratio (uPCR) | 6 months
  Change in uPCR value from baseline; expressed in mg/g.
Low density lipoprotein (LDL) | 6 months
  Change in serum LDL level from baseline; expressed in mg/dL.
Triglycerides | 6 months
  Change in serum triglycerides level from baseline; expressed in mg/dL.
Uric acid | 6 months
  Change in serum uric acid level from baseline; expressed in mg/dL.
Unfavorable disease course | 12 months
  The percentage of patients who experienced the unfavorable disease course including: glomerular disease related death; venous or arterial thromboembolic event; infection requiring hospital admission; acute kidney injury in the stage 2 or 3; sustained glomerular filtration rate reduction over 50% or initiation of kidney replacement therapy; unplanned hospital admission due to complications of nephrotic syndrome treatment.
Glomerular filtration rate | 12 months
  Change in glomerular filtration rate from baseline; expressed in mL/min/1.73m2.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Matyjek, Study Chair — Military Institute of Medicine National Research Institute
Locations (1):
- Department of Internal Diseases, Nephrology and Dialysis, Military Institute of Medicine - National Research Institute, Warsaw, Masovian District, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matyjek A, Literacki S, Niemczyk S, Rymarz A. Protein energy-wasting associated with nephrotic syndrome - the comparison of metabolic pattern in severe nephrosis to different stages of chronic kidney disease. BMC Nephrol. 2020 Aug 14;21(1):346. doi: 10.1186/s12882-020-02003-4. PMID 32795277
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Glomerular Diseases Work Group. KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases. Kidney Int. 2021 Oct;100(4S):S1-S276. doi: 10.1016/j.kint.2021.05.021. No abstract available. PMID 34556256
- [Background] Fouque D, Kalantar-Zadeh K, Kopple J, Cano N, Chauveau P, Cuppari L, Franch H, Guarnieri G, Ikizler TA, Kaysen G, Lindholm B, Massy Z, Mitch W, Pineda E, Stenvinkel P, Trevino-Becerra A, Wanner C. A proposed nomenclature and diagnostic criteria for protein-energy wasting in acute and chronic kidney disease. Kidney Int. 2008 Feb;73(4):391-8. doi: 10.1038/sj.ki.5002585. Epub 2007 Dec 19. PMID 18094682
- [Background] Kaysen GA, Gambertoglio J, Jimenez I, Jones H, Hutchison FN. Effect of dietary protein intake on albumin homeostasis in nephrotic patients. Kidney Int. 1986 Feb;29(2):572-7. doi: 10.1038/ki.1986.36. PMID 3702214
- [Background] Barsotti G, Morelli E, Cupisti A, Bertoncini P, Giovannetti S. A special, supplemented 'vegan' diet for nephrotic patients. Am J Nephrol. 1991;11(5):380-5. doi: 10.1159/000168342. PMID 1809035